CLINICAL TRIAL: NCT06211894
Title: The Effect of the Distance Between Mesh and the Urethra on Sexuality in Patients Who Underwent Transobturator Tape.
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, fatih sahin, Principal Investigator, MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: e27
Record Dates: First submitted 2023-12-27; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Urinary Incontinence; Sexual Dysfunction; Ultrasonography
Keywords: Female stress incontinence; transobturator tape; transperineal ultrasound
MeSH Terms: conditions — Urinary Incontinence; Sexual Dysfunction, Physiological | interventions — Suburethral Slings

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the urethra at the bladder neck to the nearest proximal edge of the tape: < 5 mm: Patients who achieved continence after surgery were split into two subgroups based on the distance from the posterior of the urethra at the bladder neck to the nearest proximal edge of the tape: < 5 mm and >5 mm. The position of the sling along the urethra was measured as a percentage of urethral length and referred to as the sling percentile. This measurement was calculated as follows: the proximal urethral length (distance from the sling's proximal point to the bladder neck) divided by the total urethral length (distance from the bladder neck to the external urethral meatus) on the sagittal plane, where the bladder neck and the external urethral meatus represent 0% and 100% of urethral length, respectively. Additionally, perineal ultrasound was used to evaluate various parameters including bladder descent, pubo-urethral distance, urethral thickness, detrusor thickness, cystocele descent, rectal descent, and uterine descent.
  Interventions: Procedure: transobturator tape
- the urethra at the bladder neck to the nearest proximal edge of the tape: > 5 mm: Patients who achieved continence after surgery were split into two subgroups based on the distance from the posterior of the urethra at the bladder neck to the nearest proximal edge of the tape: < 5 mm and >5 mm. The position of the sling along the urethra was measured as a percentage of urethral length and referred to as the sling percentile. This measurement was calculated as follows: the proximal urethral length (distance from the sling's proximal point to the bladder neck) divided by the total urethral length (distance from the bladder neck to the external urethral meatus) on the sagittal plane, where the bladder neck and the external urethral meatus represent 0% and 100% of urethral length, respectively. Additionally, perineal ultrasound was used to evaluate various parameters including bladder descent, pubo-urethral distance, urethral thickness, detrusor thickness, cystocele descent, rectal descent, and uterine descent.
  Interventions: Procedure: transobturator tape

INTERVENTIONS:
Procedure: transobturator tape — transobturator tape :The surgeon makes a small incision in the vagina and small incisions in the right and left groin. The surgical process is similar to the retropubic approach, but the mesh passes through the groin muscles rather than the abdominal wall. transperineal ultrasound: patients who underwent TOT and were evaluated with transperineal ultrasonography, women with incontinence 6 months after the surgery showed discrepancies in the movement of the urethra with the sling compared to continent women, along with asymmetry between the mesh arms, bladder neck descent, and varied sling positions.

SUMMARY:
Urinary incontinence, commonly observed among women aged 30 to 60, encompasses Stress Urinary Incontinence (SUI), responsible for the majority of cases. This condition significantly affects the quality of life, influencing physical, emotional, and sexual aspects. Severe cases impact libido and cause vaginal dryness, affecting not just sexual function but also relationships, leading to an overall decline in quality of life. Hence, examining sexual functions in those affected by SUI holds significance.

The study aimed to evaluate the impact of mesh-urethra distance on sexual functions using perineal ultrasound in continent patients post-transobturator tape (TOT) surgery for isolated SUI.

Patients achieving continence post-surgery were categorized based on the distance from the posterior of the urethra at the bladder neck to the nearest proximal edge of the tape: < 5 mm and > 5 mm.

Questionnaires, including the Female Sexual Function Index (FSFI) and The Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI SF), were administered preoperatively and at the 6-month postoperative follow-up.

DETAILED DESCRIPTION:
Urinary incontinence, often seen in women aged 30 to 60, involves Stress Urinary Incontinence (SUI) in most cases. It significantly affects life, impacting physical, emotional, and sexual well-being. Severe cases can lower sex drive and cause vaginal dryness, affecting not just the individual's sex life but also relationships, leading to a lower quality of life overall. That's why looking at how SUI affects sexual aspects is crucial.

The study aimed to see how the distance between the mesh and urethra after transobturator tape (TOT) surgery might affect sexual function in patients who no longer experienced incontinence. Patients were divided based on this distance, and surveys like the Female Sexual Function Index (FSFI) and The Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI SF) were used before and six months after surgery.

ELIGIBILITY:
Inclusion Criteria:

-Continent patients ages 18 to 45 who underwent mid-urethral sling (MUS) surgery due to isolated SUI were included in the study

Exclusion Criteria:

* Patients who experienced surgical failure in incontinence surgery,
* who had undergone previous vaginal surgeries, who had a history of hysterectomy,
* who underwent additional surgeries during the same session,
* who had pelvic organ prolapse, who had received radiation therapy,
* who had a diagnosis of malignancy,
* who were menopausal, who received external hormone treatment,
* who were sexually inactive, whose partners had erectile dysfunction,
* who did not attend postoperative follow-up appointments,
* who became postoperatively pregnant,
* who had undergone non-synthetic mesh (autologous fascia) surgery for SUI were excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Between January 2020 and January 2022, a total of 82 continent patients ages 18 to 45 who underwent MUS surgery due to isolated SUI were included in the study
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the significance of postoperative FSFI scores on sexual functions in patients with continent status who underwent TOT surgery due to isolated SUI. | 6 months
  The primary outcome measure involves assessing the impact of postoperative FSFI (Female Sexual Function Index) scores specifically on the sexual functions of patients who have maintained continence status and underwent TOT (Transobturator Tape) surgery attributable to isolated Stress Urinary Incontinence (SUI)
To assess the significance of sexual functions using The ICIQ-UI SF score in patients with continence status who underwent TOT surgery due to isolated SUI. | 6 months
  evaluating the relevance of sexual functions utilizing The ICIQ-UI SF (International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form) score among patients maintaining continence status following Transobturator Tape (TOT) surgery due to isolated Stress Urinary Incontinence (SUI)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Cemil Tascıoglu City Hospital, Istanbul
  - Prof.Dr.Cemil Taşcıoğlu Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No